CLINICAL TRIAL: NCT03023683
Title: U19 Influenza Immunity: Protective Mechanisms Against a Pandemic Respiratory Virus. Project 1: B-cell Immunity to Influenza
Brief Title: Protective Mechanisms Against a Pandemic Respiratory Virus (SLVP024)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-24965; U19AI057229-07 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2017-01

CONDITIONS: Influenza
Keywords: Live, attenuated influenza vaccine; Children and young adults
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: 2-8 yo healthy non-twins (Other): Participants will be given seasonal live, attenuated influenza vaccine (LAIV), FluMist® . Children with no prior influenza vaccine history will receive a second dose of LAIV at least 28 days after the first study dose.
  Interventions: Biological: FluMist®
- Group B: 18-49 yo healthy non-twins (Other): Participants will be given seasonal LAIV, FluMist® .
  Interventions: Biological: FluMist®

INTERVENTIONS:
Biological: FluMist® — Influenza Virus Vaccine Live, Intranasal Spray

SUMMARY:
The purpose of the study is to investigate and compare the human immune response in epithelial cells of the nasopharyngeal mucosa and in blood to live, attenuated influenza vaccine (LAIV) in adults and in children.

DETAILED DESCRIPTION:
The objective of the protocol is to investigate the human innate and adaptive immune responses in blood (only for adults) and nasopharyngeal mucosa resident cells to the live, attenuated influenza vaccine (LAIV) in both adults and children. The investigators hope to learn how the upper respiratory tract (URT) epithelial cells, the primary target of respiratory viruses, and the B cells and T cells, two major components of the immune system, respond to the influenza vaccine.

The volunteers will be enrolled in two age groups:

Group A: Up to 12 healthy non-twin volunteers, 2-8 years old, will be given seasonal LAIV. Each volunteer will complete a total of 3 visits. Volunteers will be divided in 2 sub-groups A-1 (n=6) and A-2 (n= 6) in order to collect nasopharyngeal swabs on different schedules (Day 1 or Day 2). Volunteers will be assigned to these sub-groups based on convenience sampling. Both sub-groups will complete the Day 0 and Day 28 visits and one visit at either Day 1 or Day 2 post-immunization. Specimens will include nasopharyngeal swabs collected at Day 1 for Sub-group A1 and Day 2 for Sub-group A-2, and Day 28 for both sub-groups. No blood samples will be collected in this age group.

Children with no prior influenza vaccine history will receive a second dose of vaccine (LAIV) at least 28 days after the first study dose, according to the ACIP guidelines.

Group B: Up to 18 healthy non-twin volunteers, 18-49 yrs old, will be given seasonal LAIV vaccine. Each volunteer will complete a total of 5 visits. Volunteers will be divided into 3 sub-groups B-1, B-2 and B-3 in order to collect nasopharyngeal swabs and blood specimens on different schedules (Day 0-6 hrs, Day 1 or Day 2). Volunteers will be assigned to these sub-groups based on convenience sampling. All sub-groups will complete visits at Day -7, Day 0 pre-immunization, Day 7 and Day 28 and 1 additional time point: Sub-group B-1 at Day 0, 6 hours post-immunization, Sub-group B-2 at Day 1 and Sub-group B-3 at Day 2. A nasopharyngeal swab will be collected at each visit except for Day 0 (baseline) and Day 7. A blood sample will be collected at each visit except Day -7

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, ambulatory 2-8 years old (Group A) or 18-49 years old (Group B).
2. Willing to complete the informed consent process (including assent for minors 7 years old and above).
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history by review of inclusion and exclusion criteria and vital signs.

Exclusion Criteria:

1. Prior off-study vaccination with the current 2012-2013 seasonal TIV or LAIV.
2. Allergy to egg or egg products, or to vaccine components, including gentamicin, gelatin, arginine or MSG (LAIV)
3. Life-threatening reactions to previous influenza vaccinations
4. Asthma or history of wheezing
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Blood pressure >150 systolic or >95 diastolic at the first study visit and on the day of vaccination.
9. Hospitalization in the past year for congestive heart failure or emphysema.
10. Chronic Hepatitis B or C.
11. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible)
12. Participants in close contact with anyone who has a severely weakened immune system should not receive LAIV
13. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
14. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
15. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
16. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
17. Receipt of blood or blood products within the past 6 months or planned used during the study.
18. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
19. Receipt of Inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last visit ( Day ~28 after study vaccination)
20. Receipt of live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last visit (Day ~28 after study vaccination)
21. Need for allergy immunization (that cannot be postponed) during the study period.
22. History of Guillain-Barré syndrome
23. Pregnant or lactating woman (NA for children in Group A)
24. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
25. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned donation prior to completion of the last visit.
26. A current member of the clinical study team.
27. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 2 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Harry Greenberg, MD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A: 2-8 yo Healthy Non-twins | Group B: 18-49 yo Healthy Non-twins
Started | 0 | 18
Completed | 0 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 2-8 yo Healthy Non-twins | Group B: 18-49 yo Healthy Non-twins | Total
Number analyzed (Participants) | 0 | 18 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 28.07 (8.09) | 28.07 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 7 | 7
  Male |  | 11 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 18 | 18
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 5 | 5
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 10 | 10
  More than one race |  | 3 | 3
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 18 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Each Arm Who Received Influenza Vaccine
Time Frame: Day 0 to 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 2-8 yo Healthy Non-twins | Group B: 18-49 yo Healthy Non-twins
Number analyzed (Participants) | 0 | 18
Participants | 0 | 17

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 2-8 yo Healthy Non-twins | Group B: 18-49 yo Healthy Non-twins
Number analyzed (Participants) | 0 | 17
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 28
Description: Clinical Assessment performed at each visit
Arm/Group | Group A: 2-8 yo Healthy Non-twins | Group B: 18-49 yo Healthy Non-twins
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/17
Other Adverse Events (participants affected / at risk) | 0/0 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No